CLINICAL TRIAL: NCT05102721
Title: A Phase 1b/2 Trial of Immunotherapy With Avelumab and Pepinemab As Second Line For Patients With Metastatic Pancreatic Adenocarcinoma
Brief Title: Trial of Immunotherapy With Avelumab and Pepinemab As Second Line For Patients With Metastatic Pancreatic Adenocarcinoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vaccinex Inc. (Industry)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SGIP21027
Record Dates: First submitted 2021-10-21; First posted 2021-11-01 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
Keywords: Metastatic Pancreatic Adenocarcinoma
MeSH Terms: interventions — avelumab; pepinemab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): Single arm, all patients serially enrolled to combination doses of Avelumab and Pepinemab
  Interventions: Drug: Avelumab and Pepinemab

INTERVENTIONS:
Drug: Avelumab and Pepinemab — IV Infusions every two weeks.

SUMMARY:
This trial will assess the safety and tolerability of Pepinemab in combination with Avelumab in patients with metastatic pancreatic adenocarcinoma that has progressed after first line chemotherapy. Phase 2 will assess the efficacy of this combination therapy.

DETAILED DESCRIPTION:
Pancreatic adenocarcinoma (PDAC) is the third leading cause of cancer related deaths with an incidence expected to increase over the next decade.3 Despite modest advances in conventional chemotherapy, five-year survival remains dismal at 5-10%.4 Therefore, the development of effective therapies for treating PDAC represents a significant unmet medical need. The near 95% 5 year mortality observed in PDAC is in part due to advanced disease stage at presentation, and a propensity for recurrence following curative intent resection. As a result, 5FU regimens (including FOLFIRINOX) or Gemcitabine based cytotoxic chemotherapies are standard of care for patients who present with both resectable and unresectable disease.5,6 However, despite advances in cytotoxic chemotherapy, a majority of patients fail to respond to first line therapy, and only around 10-15% of patients experience treatment response in the second line setting, while a third of patients experience grade 2-3 toxicities from second-line regimens.7,8 Thus, novel second-line treatments with improved toxicity profiles compared to cytotoxic chemotherapy are a dire medical need and strongly supported by patient advocates of this dismal disease.

A body of clinical and preclinical work has shown that the profoundly immunosuppressive tumor microenvironment (TME) in PDAC remains a significant barrier to effective cytotoxic and immune based therapies.9-11 Somewhat unique to PDAC, a dense fibrotic stroma is infiltrated with bone-marrow derived myeloid cells of monocytic and granulocytic origin including tumor associated macrophages (TAM) neutrophils (TAN) and immature suppressive myeloid progenitors (MDSCs). Tumor-infiltrating myeloid cells are highly immunosuppressive and the most prevalent immune cells found in the TME of PDAC.12,13 These cells produce immunosuppressive cytokines (Il6, Il10, Il4), secrete considerable amounts of arginase, and produce reactive oxygen species, essentially shielding the tumor from effective T cell immunity.14 Thus, PDAC is an immunologically "cold" tumor with minimal T cell adaptive response, which in part explains the failure of immune-checkpoint blockade therapy to demonstrate efficacy in PDAC.15-17 Previous work has shown that small molecule chemokine inhibitors targeted at monocytic myeloid cells (TAM precursors) can effectively prevent mobilization and trafficking of these cells to the TME, and improve the standard of care chemotherapy in both preclinical and clinical studies (NCT01413022, NCT02732938, NCT02345408).18 However, these successes in reprogramming of the tumor microenvironment are accompanied by a compensatory increase in immunosuppressive granulocytes (TANs and pmn-MDSCs), resulting in treatment resistance to single subtype myeloid blockade.18 Based on this finding of myeloid compensation by TANs in the absence of TAMs, and the potential therapeutic value in dual myeloid inhibition, new therapies targeted at both myeloid subtypes represent a unique opportunity for exposing PDAC to effective immune surveillance.13,19 Human data has previously correlated both SEMA4D and Plexin B1 expression with nodal metastasis, invasiveness, and worse overall survival in patients who underwent resection for PDAC.25 Analysis of resected tumor specimens demonstrate an avid infiltrate of Semaphorin 4D cells (Figure 3B). Concomitantly, myeloid suppressor cells within the PDAC TME demonstrate avid expression of Semaphorin 4D receptors, Plexin B1 and Plexin B2 (Figure 3B). Thus, Semaphorin 4D blockade represents a novel immunotherapeutic strategy within the PDAC TME.

The trial is carried out in two stages. In Phase 1b, a maximum number of up to 44 patients is accrued, but as few as 16 patients are needed and 1000 simulations of this model anticipates between 24-29 patients. Phase 1b will continue until 16 evaluable patients accrue in a dose. Once 16 patients have accrued to a particular dose based on the BOIN design, the MTD dose is established as the dose yielding 30% or lower DLT rate. If there is 1 or less objective responses among these 16 patients, the study will be stopped early for efficacy futility according to Simon's two-stage design.1,2 If after evaluation of futility the trial is meeting early markers of efficacy (at least 2/16 responses), an expansion cohort will begin. Dose escalation will cease and all patients will subsequently enter the second stage of the trial at the MTD dose defined by Phase 1b. In this expansion cohort, Phase 2, up to 24 patients will be enrolled. These patients will be followed for objective response rates by RECIST 1.1 criteria and iRECIST. When combined with the 16 patients from Phase 1b, the Phase 2 cohort will total an evaluable sample size of 40. If there are 5 or more responses among these 40 patients, we reject the null hypothesis and claim that the treatment is promising. An objective response rate of 23% will afford a 10% type 1 error with 80% power to detect a difference. The null hypothesis is that the true response rate is 0.10 or less, and the alternative hypothesis is that the true response rate is 0.23 or greater. The design controls the type I error rate at 0.1 and yields the power of 0.8.

ELIGIBILITY:
Inclusion Criteria:

* Patient or legally acceptable representative must be able to understand and willing to sign an IRB approved written informed consent document.
* Patients must be 18 years or older
* Patients must have histologically confirmed metastatic pancreatic adenocarcinoma.
* Patients must have radiographically measurable disease defined as non-radiated lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as greater than or equal to 10mm with calipers by radiographic exam.Further details listed in section 5.5.
* Patients must have received 5FU or Gemcitabine based first line treatment (in combination with platinum, topoisomerase I inhibitor, or nab-paclitaxol) for metastatic disease with evidence of treatment failure or intolerance.
* If a subject received therapy in the adjuvant/neoadjuvant setting:
* Tumor recurrence must have occurred no sooner than 6 months after completion of the last dose of therapy.
* Radiation therapy for the locally advanced disease is allowed
* The patient must have a life expectancy of minimum 3 months.
* Patient must have normal bone marrow and organ function as defined below:

  * Absolute neutrophil count >1,500/mcl
  * Platelets >100,000/mcl
  * Hemoglobin >9.0 g/dL
  * Creatinine should be below the upper limit of normal OR
  * Creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Patient not on anticoagulation must have international Normalized Ratio (INR) and activated partial thromboplastin time (PTT) <1.5 upper limit of normal.
* Patient will have an ECOG performance status of 0, 1, or 2
* Patient must consent for baseline and on treatment biopsies, if prior baseline biopsies have been performed, and stored within the University of Rochester Cancer Library, then baseline biopsies are not necessary. Baseline biopsy must be of a lesion post-relapse.
* Patients with biliary stents for obstruction may be included in the study
* Female subjects of childbearing potential must demonstrate a negative urine or serum pregnancy test.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of the study treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Male subjects with a female partner of child-bearing potential must agree to use 2 adequate methods of contraception (barrier + hormonal for example).

Exclusion Criteria:

* Patient with any histologic variant of PDAC such as adenosquamous, acinar cell, duodenal adenocarcinoma, or ampullary adenocarcinoma
* Patient has a history of other malignancy ≤ 3 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix.
* Patient who is receiving or has received an investigational immunotherapy, investigational combinations of cytotoxic chemotherapy such as liposomal irinotecan are permitted
* Patient has a history of allergic reactions attributed to compounds of similar chemical or biologic composition to Pepinemab (VX15/2503) or Avelumab
* Patient with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, any clinically active malabsorption syndrome, inflammatory bowel disease, any condition that increases the risk of severe irinotecan gastrointestinal toxicity, or psychiatric illness/social situations that would limit compliance with study requirements
* Has an active autoimmune disease, or a documented history of autoimmune disease or a syndrome that requires steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be exceptions to this rule.
* Has had an allogenic tissue/solid organ transplant.
* Has interstitial lung disease or a history of pneumonitis that required oral or intravenous glucocorticoids to assist with management.
* Has received or will receive a live vaccine within 30 days prior to the first administration of study medication. Flu vaccines that do not contain live virus are permitted.
* Has known active Hepatitis B or C.
* Patient who is pregnant and/or breastfeeding.
* Persisting toxicity related to prior anti-cancer therapy
* Major surgery or use of investigational drug within the 28 days before the start of treatment
* Current alcohol or drug abuse
* Prior organ or bone marrow transplantation
* Inability to comply with visit schedule or other protocol requirements including mandatory study biopsies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-12-10 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 10 years
  Measured by adverse event severity and quantity

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Mulkerin, MD, Principal Investigator — WCICTOResearch@urmc.rochester.edu
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
A complete and final study protocol will be made publicly available through the University of Rochester Cancer Center Community Oncology Research Program Research Base Protocol and Data Sharing Committee. The full protocol and data will be made publicly available no later than the publication date of the study findings from the final dataset. The protocol will include a detailed description of the study population, hypotheses tested, measurement and assessment information, data definitions and codes, and the analysis plan utilized. We will be collecting identifying information. The final dataset will be stripped of identifiers prior to release for sharing. Published papers will be made available in portable document format.
Time Frame: The data will be available for 7 years from accrual of the first subject